CLINICAL TRIAL: NCT06792175
Title: Mental Health, Intellectual and Neurodevelopmental Disorder Detection With Artificial Intelligence Models: Testing Speech-Based Machine Learning Algorithms for Clinical Assessment and Risk Stratification in Mental Health Presentations
Brief Title: Mental Health, Intellectual and Neurodevelopmental Disorder Detection With Artificial Intelligence Models
Acronym: MINDAIM
Status: Enrolling by invitation | Type: Observational
Sponsor: Psyrin Inc. (Industry)
Collaborators: Allwell Behavioral Health Services (Unknown); The Brookline Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: PSYRIN-0004
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-02

CONDITIONS: Autism Spectrum Disorder; Depression - Major Depressive Disorder; Anxiety, Generalized; Bipolar Disorder (BD); Attention Deficit Hyperactivity Disorder (ADHD); Schizophrenia Spectrum &Amp; Other Psychotic Disorders; Post Traumatic Stress Disorder; Obsessive Compulsive Disorder (OCD)
Keywords: Artificial Intelligence; Natural Language Processing; Acoustic Analysis; Acoustic Biomarkers; Clinical Testing; Vocal Biomarkers; Machine Learning; Mental Health; Speech Analysis
MeSH Terms: conditions — Autism Spectrum Disorder; Generalized Anxiety Disorder; Bipolar Disorder; Attention Deficit Disorder with Hyperactivity; Stress Disorders, Post-Traumatic; Obsessive-Compulsive Disorder; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Audio of speech collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Solicue (Any Mental Health Disorder): Any participant enrolled in the study and not part of additional analysis group.
  Interventions: Diagnostic Test: Solicue Machine Learning Models
- Solicue & Mercuria (Bipolar Disorder & Major Depressive Disorder): Any participant enrolled in the study and exhibiting depressive symptoms as measured by PHQ-9 score.
  Interventions: Diagnostic Test: Solicue Machine Learning Models; Diagnostic Test: Mercuria Machine Learning Models

INTERVENTIONS:
Diagnostic Test: Solicue Machine Learning Models — A comprehensive machine-learning tool aimed at providing probability estimates for several compatible disorders, including Attention Deficit Hyperactivity Disorder (ADHD), Autism Spectrum Disorder (ASD), Bipolar Affective Disorder (BPAD), Generalized Anxiety Disorder (GAD), Major Depressive Disorder (MDD), Obsessive Compulsive Disorder (OCD), Post-Traumatic Stress Disorder (PTSD), and Schizophrenia Spectrum Disorders (SSD). By offering a multi-diagnostic assessment based on speech analysis, Solicue aims to assist clinicians in navigating this complexity and potentially identifying conditions that might otherwise be overlooked in initial assessments.
  Solicue leverages machine learning to analyze a wide range of clinically relevant speech features, including linguistic content, prosodic elements (such as pitch, rhythm, and intonation), and other paralinguistic features.
  Other Names: Solicue; Psyrin Speech Analysis; Solicue Artificial Intelligence
Diagnostic Test: Mercuria Machine Learning Models — Mercuria is designed to stratify the risk of bipolar disorder in individuals presenting with depressive symptoms. This is a critical clinical need, as misdiagnosis of bipolar disorder as unipolar depression is common and can lead to inappropriate treatment, potentially worsening outcomes. By analyzing speech patterns characteristic of bipolar disorder, Mercuria aims to provide an additional tool for clinicians to differentiate between these conditions more accurately, guiding appropriate treatment decisions.
  Mercuria leverages machine learning to analyze a wide range of clinically relevant speech features, including linguistic content, prosodic elements (such as pitch, rhythm, and intonation), and other paralinguistic features.
  Other Names: Mercuria; Mercuria Artificial Intelligence
  Groups: Solicue & Mercuria (Bipolar Disorder & Major Depressive Disorder)

SUMMARY:
This study investigates whether AI-driven analysis of speech can accurately predict clinical diagnoses and assess risk for various mental or behavioral health conditions, including attention-deficit/hyperactivity disorder (ADHD), autism spectrum disorder, bipolar disorder, generalized anxiety disorder, major depressive disorder, obsessive compulsive disorder (OCD), post-traumatic stress disorder (PTSD), and schizophrenia. We aim to develop tools that can support clinicians in making more accurate and efficient diagnoses.

ELIGIBILITY:
Inclusion Criteria

1. Participants aged between 16 and 60 years.
2. Individuals currently undergoing or referred for clinical assessment of mental or behavioral health conditions (including but not limited to ADHD, ASD, BPAD, GAD, MDD, OCD, PTSD, SSD)
3. Fluent in English
4. Capable of providing informed consent, or in the case of minors, having a parent or legal guardian who can provide consent on their behalf.
5. Access to a device (smartphone, tablet, or computer) with a microphone and stable internet connectivity, necessary for completing the speech tasks.

Exclusion Criteria

1. Individuals experiencing acute mental health crises or severe symptoms that would preclude meaningful participation in the study, including acute intoxication.
2. Severe cognitive impairment or intellectual disability that would prevent understanding of the study procedures or completion of the speech tasks.
3. Lack of fluency in English.
4. Technical limitations: Inability to access a suitable device or internet connection for completing the speech tasks

Ages: 13 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: The MIND AIM study aims to recruit a diverse and representative sample of individuals seeking mental health assessments in various clinical settings. This broad inclusion criteria ensures high ecological validity, capturing the wide range of presentations and comorbidities commonly encountered in real-world mental health practice.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Speech Battery ("PSY-10") audio | At initial assessment
  The speech battery consists of prompt-based tasks designed to elicit speech responses from participants in the form of monologues. This includes text reading, recall, and picture description tasks.
Clinical diagnosis | 0 months, 3 months, 6 months
  Clinician diagnosis will be recorded for each participant at first assessment, 3-month, and 6-month follow-up. Diagnoses will be made according to ICD-11 or DSM-5 criteria for the compatible disorders: ADHD, ASD, BPAD, GAD, MDD, OCD, PTSD, and SSD. Additional relevant labels such as other mental health disorders, clinical high risk (CHR) and substance use may be recorded.
Performance of AI models | 0 months, 3 months, 6 months
  The performance of the Mercuria and Solicue AI models will be evaluated using performance metrics of accuracy, balanced accuracy, sensitivity (recall), specificity, positive predictive value (precision), negative predictive value, F1 score, AUC-ROC. Predicted labels will be compared with the ground truth clinical diagnoses obtained from the participating mental health clinics. Confidence acceptance threshold will be set.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | At initial assessment
  The PHQ-9 is a 9-item self-reported questionnaire that assesses the severity of depressive symptoms.
Mood Disorder Questionnaire (MDQ) | At initial assessment
  The MDQ is a 15-item self-report screening instrument designed to detect bipolar spectrum disorders. It consists of 13 yes/no questions about manic symptoms, followed by two questions about the co-occurrence and impact of these symptoms.
DSM-5 Level 1 Cross-Cutting Symptom Measure (DSM-XC) | At initial assessment
  The DSM-5 Level 1 Cross-Cutting Symptom Measure is a 23-item self-report questionnaire that screens for 13 psychiatric domains, including depression, anxiety, and substance use.
Reported Distress | After initial assessment
  To assess the safety of online speech assessment during clinical evaluation at initial intake. The safety of online speech assessment will be measured by severity of reported distress measured using the User Feedback Form (UFF).

CONTACTS AND LOCATIONS:
Overall Officials: Julianna Olah, B.Sc., M.A., M.Sc., Ph.D., Principal Investigator — Psyrin Inc.; Atta-ul Raheem R Chaudhry, B.Sc. (Hons.), M.B.B.S., Principal Investigator — Psyrin Inc.
Locations (2):
- United States (2):
  - The Brookline Center, Brookline, Massachusetts
  - Allwell Behavioral Health Services, Zanesville, Ohio

IPD SHARING:
Plan to Share IPD: Undecided